CLINICAL TRIAL: NCT05728268
Title: Neoadjuvant Dose-dense Chemotherapy for HR+/HER2- Breast Cancer Patients With High Proliferation Index
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shantou Central Hospital (Other)
Collaborators: Shantou University Medical College (Other); Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Wu, Dr., Shantou Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShantouCH02
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose-dense arm (Experimental)
  Interventions: Drug: dose-dense nab-paclitaxel followed by EC

INTERVENTIONS:
Drug: dose-dense nab-paclitaxel followed by EC — dose-dense nab-paclitaxel followed by EC

SUMMARY:
Studies have shown that dose-dense chemotherapy reduces the risk of recurrence and death of breast cancer patients comparing with standard-schedule chemotherapy. But some research data indicate that HR+/HER2- breast cancer patients benefit from dose-dense chemotherapy while some have negative results. How to identify HR+/HER2 breast cancer patients who are more likely to benefit from dose-dense chemotherapy is strongly necessary. Ki67 is a marker reflecting the proliferation of tumor cells. Breast cancer patients with high Ki67 are more likely to benefit from dose-dense chemotherapy. The purpose of this project is to investigate the efficacy and safety of neoadjuvant dose-dense chemotherapy for HR+/HER2- breast cancer patients with high proliferation index. At the same time, we will explore biomarkers, such as MammaPrint and BluePrint, to further identify patients who benefit more from neoadjuvant dose-dense chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Females with age of 18 to 70 years old.
* Newly diagnosed breast cancer patients.
* Planned neoadjuvant chemotherapy.
* Hormone receptor status: Estrogen receptor (ER)-positive or Progesterone Receptor (PR)- positive.
* HER2/neu-negative.
* Ki67≥30%.
* Clinical stage IIB-IIIC.
* Informed consent form understood and signed.
* Patient agrees to all follow-up visits.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Women of childbearing potential must have a negative serum pregnancy test.

Exclusion Criteria:

* Metastatic disease
* Pregnancy.
* Nursing mothers.
* Active or uncontrolled infection.
* Presence of another malignancies.
* Granulocyte count < 1.5*10^9/L.
* Platelet count < 100*10^9/L.
* Hemoglobin < 90g/L.
* Serum Creatinine more than 1.5 upper limit.
* AST and ALT more than 2.5 upper limit.
* LVEF< 50%.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
RCB | 7 days
  Residual Cancer Burden

CONTACTS AND LOCATIONS:
Locations (1):
- Shantou Central Hospital, Shantou, Guangdong, China